CLINICAL TRIAL: NCT01945931
Title: Evaluation of a Smartphone Application to Reduce Adverse Pregnancy Outcomes in Ethiopia: A Cluster-randomised Controlled Trial
Brief Title: Evaluation of a Smartphone Application to Reduce Adverse Pregnancy Outcomes in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Stine Lund, MD, PhD fellow, MD, PhD fellow, University of Copenhagen
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SafeDeliveryApp
Record Dates: First submitted 2013-09-05; First posted 2013-09-19 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Maternal Mortality; Perinatal Mortality
Keywords: Maternal health; perinatal health; mHealth; smartphone; mobile phone; Ethiopia
MeSH Terms: conditions — Maternal Death; Perinatal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Safe Delivery Smartphone Application (Experimental): The safe delivery smartphone application is designed to train midwives and other birth attendants in developing countries in management of normal and complicated deliveries. The safe delivery smartphone application will be introduced to health workers in the intervention clusters.
  Interventions: Other: Safe Delivery Smartphone Application
- Control (No Intervention): Health workers in the control clusters will not have access to the Safe Delivery App

INTERVENTIONS:
Other: Safe Delivery Smartphone Application — The safe delivery smartphone application is designed to train midwives and other birth attendants in developing countries in management of normal and complicated deliveries. The application is furthermore intended as a reference tool that could be used during clinical work for example for preparation before attending a birth, in a situation when a complication occurs, or for debriefing and self-evaluation after a complication. The application features four animated videos with clinical instructions of 3-8 minutes duration and written lists of essential obstetric drugs (indications, contraindications, dosage and administration and side effects) and essential equipment for a safe delivery.
  Arms: Safe Delivery Smartphone Application

SUMMARY:
The purpose of this trial is to determine if the safe delivery smartphone application distributed to health workers in Ethiopia will decrease perinatal mortality and the incidence of postpartum haemorrhage. It is also the purpose to determine if the safe delivery smartphone application distributed to health workers in Ethiopia will increase health workers knowledge and skills in intra-partum management of active management of third stage labour 2) treatment of post-partum haemorrhage 3) manual removal of placenta and 4) neonatal resuscitation.

DETAILED DESCRIPTION:
Abstract Hypothesis A safe delivery smartphone application distributed to health workers in Ethiopia will decrease perinatal mortality and the incidence of postpartum haemorrhage

A safe delivery smartphone application distributed to health workers in Ethiopia will increase health workers knowledge and skills in intra-partum management of active management of third stage labour 2) treatment of post-partum haemorrhage 3) manual removal of placenta and 4) neonatal resuscitation

Intervention A safe delivery smartphone application with animated videos to improve clinical management during delivery will be introduced in the intervention clusters

Design Cluster randomized controlled trial with health facilities as the unit of randomization

Area Nole Kaba, Haru, Homa, Genji and Gimbie districts in Ethiopia

Population Pregnant women and their newborns delivered in a randomized health facility. For secondary outcomes health workers at randomized health facilities.

Sample size 77 health facilities with minimum 2 health workers per facility and 30 deliveries per health worker

Duration Pregnant women will be enrolled at delivery and followed to 7 days postpartum

Outcomes Primary outcomes are perinatal mortality and postpartum haemorrhage. Secondary outcomes are health workers knowledge and skills

Study time Data collection expected from September 2013 to September 2014

ELIGIBILITY:
Inclusion Criteria:

• Women in active labor

Exclusion Criteria:

• None

Ages: 10 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3601 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Perinatal mortality (stillbirth and early neonatal death) | Participants will be followed from delivery until 7 days postpartum
Postpartum haemorrhage | Participants will be followed from delivery until two hours postpartum

SECONDARY OUTCOMES:
Health workers clinical performance in active management of third stage of labour, postpartum haemorrhage and manual removal of placenta | 0, 6 and 12 months
Health workers clinical performance in management of neonatal resuscitation | 0, 6 and 12 months
Health workers knowledge of management of active management of third stage of labour, manual removal of placenta and postpartum haemorrhage | 0, 6 and 12 months
Health workers knowledge of management of neonatal resuscitation | 0, 6 and 12 months

OTHER OUTCOMES:
Mortality stratified according to gestational age and birth weight | Participants will be followed from delivery until 7 days postpartum
Use of the Safe Delivery application (when, how much and by whom) | Participants will be followed during the 12 months trial period
Process indicators of services provided | Participants will be followed from delivery until 7 days postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, København V, Denmark

REFERENCES:
- [Derived] Christiansen AH, Sorensen BL, Boas IM, Bedesa T, Fekede W, Nielsen HS, Lund S. The impact of the Safe Delivery Application on knowledge and skills managing postpartum haemorrhage in a low resource setting: a cluster randomized controlled trial in West Wollega region, Ethiopia. Reprod Health. 2023 Jun 16;20(1):91. doi: 10.1186/s12978-023-01635-7. PMID 37328731
- [Derived] Lund S, Boas IM, Bedesa T, Fekede W, Nielsen HS, Sorensen BL. Association Between the Safe Delivery App and Quality of Care and Perinatal Survival in Ethiopia: A Randomized Clinical Trial. JAMA Pediatr. 2016 Aug 1;170(8):765-71. doi: 10.1001/jamapediatrics.2016.0687. PMID 27322089